CLINICAL TRIAL: NCT05235191
Title: A Randomized Controlled Trial Study to Assess the Effectiveness and Safety of Methadone Versus Placebo for the Control of Neuropathic Pain in Different Etiologies
Brief Title: Effectiveness and Safety of Methadone Versus Placebo for the Control of Neuropathic Pain in Different Etiologies
Acronym: METHA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Daniel Ciampi Araujo de Andrade, MD, PhD, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 45397515.2.0000.0068
Record Dates: First submitted 2020-06-18; First posted 2022-02-11 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Neuropathic Pain
Keywords: Methadone; Neuropathic Pain; Opioid; Pain
MeSH Terms: conditions — Neuralgia; Pain | interventions — Methadone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- methadone (Experimental): In this arm patients will take methadone 5mg
  Interventions: Drug: methadone tablets
- placebo (Placebo Comparator): In this arm patients will take placebo tablets (the same number, color and physical aspects as the methadone tablets).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: methadone tablets — The intervention with the active drug (methadone) will start with the dose of 1 tablet (5 mg) twice a day (every 12 hours) and titrated on subsequent visits up to the maximum dose of 6 tablets a day (totaling 30 mg divided into 2 daily doses to facilitate therapeutic adherence).
  Other Names: Mytedom
  Arms: methadone
Drug: Placebo — In this arm patients will take placebo tablets (the same number, color and physical aspects as the methadone tablets).
  Arms: placebo

SUMMARY:
Opioids are currently ranked as third-line agents for neuropathic pain (NP) treatment. The opioids more frequently tested for NP were tramadol, oxycodone and morphine. In the present study test the safety and effectiveness of methadone in patients with NP who remain symptomatic despite the use of first and second line drugs in a placebo-controlled randomized approach.

DETAILED DESCRIPTION:
Background: neuropathic pain (NP) is highly refractory and it is estimated that about 40% of patients remain symptomatic despite the use of first and second line drugs. Opioids are currently ranked as third-line agents for NP treatment. The opioids more frequently tested for NP were tramadol, oxycodone and morphine. In the present study test the effectiveness and safety of methadone, an opioid agonist and glutamate n-methyl-d-aspartate (NMDA) receptor antagonist in patients with NP who remain symptomatic despite the use of first and second line drugs in a placebo-controlled randomized approach.

Patients and Methods: this is a randomized, placebo controlled superiority trial including 80 subjects, aged between 18 and 85 years, with NP, that will be randomized to receive methadone or placebo in a 1:1 ratio. Enrollment will take place at the Pain Center of the University of São Paulo and it will include patients from primary care clinics from an area of 2 million people addressed to specialized care at a referral center.

Expected results: the study hypothesis is that methadone is superior to placebo and it is safe to use that medication in patients with neuropathic pain.

Recruitment time will be extended by 12 months due to dropouts related to the Covid pandemic. We have had dropouts due to a few patients developing covid and also due to patients having fear to become infected while attending hospital visits

ELIGIBILITY:
Inclusion Criteria:

1. Presence of an exclusive neuropathic pain (without other main pain syndrome occurring concomitantly at the same body area);
2. Pain lasting at least 6 months (chronic) and being present most of the days;
3. Pain fulfilling the current IASP (The International Association for the Study of Pain) criteria for defined Neuropathic Pain and with a score on the DN4 questionnaire (Douleur Neuropathique Pain 4 Questions) ≥ 4 (positive);
4. The pain must be of at least moderate intensity (score on a visual analogue pain scale ≥ 40/100) despite the use of first and second line drugs in an adequate dosing.

Exclusion Criteria:

* Patients under the age of 18 or over 85;
* Who has neuropathic pain duration less than 6 months;
* Who do not have an exclusive neuropathic pain (without other main pain syndrome occurring concomitantly at the same body area);
* Patients with neuropathic pain intensity less than 40 out of 100 on a visual analogue pain scale;
* Who scored less than 4 on the DN4 scale;
* Who wishes at any time to abandon the study;
* Patients with a previous allergic reaction to any of the drugs involved in the study (methadone) or placebo components;
* Patients in current use or in the last 14 days of medication (s) inhibitor (s) of monoamine oxidase (MAOI) or other medications with potential drug interaction with methadone;
* Patients in current continuous use of opioids (including methadone);
* Patients with a history of opioid abuse;
* Patients with a history of heavy/abusive alcohol consumption;
* Who is under judicial litigation, police custody or institutionalized for other reasons;
* Pregnant women, lactating women or women of childbearing age (without the use of an adequate contraceptive method);
* Patients with participation in another research protocol that implies the use of some medication during the 30 days preceding the inclusion in the project;
* Who uses illegal drugs;
* Patients unable to assess the risks and benefits of participating in the present study (eg, language barriers, psychiatric disorders or cognitive impairment);
* The presence of psychiatric disorders such as uncontrolled posttraumatic stress disorder, uncontrolled depression, uncontrolled anxiety disorder and suicidal ideation;
* Who has acute or chronic renal failure;
* Who has liver or heart failure;
* Who has a history of elevated cardiac QT interval, risk factors for elevated QT interval (including drugs that can prolong that interval), as well as cardiac arrhythmias/cardiac conduction abnormalities;
* Who has serious or intolerable adverse reactions to any component of the drugs involved in the study;
* Patients with a previous history of severe asthma or severe respiratory disease that may increase the risk of respiratory failure;
* Patients with active infectious gastrointestinal disease, active inflammatory gastrointestinal disease and obstruction of the gastrointestinal tract;
* Patients with history of recent traumatic brain injury (less than 7 days) or severe at any time interval;
* Who has moderate or severe obstructive sleep apnea-hypopnea syndrome;
* Who has uncontrolled hypothyroidism or hyperthyroidism;
* Patients with a history of uncontrolled epilepsy;
* Patients with current intracranial hypertension;
* Patients with grade III obesity (BMI ≥ 40 kg / m2).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Pain intensity change from baseline, assessed by the visual analogue scale (VAS) | 0 and 56 days
  To evaluate the analgesic effect of methadone (number of patients with ≥ 30% pain intensity change from baseline) compared to placebo in patients with neuropathic pain (NP) of different etiologies.
  The impact on the average change in the intensity of NP (baseline) will be evaluated, with the main objective being a higher number of responders in the methadone at study completion compared to the placebo group. Responder is defined as pain intensity reduction greater than or equal to 30% compared to the baseline intensity of NP. It will be measured according to a visual analogue scale (VAS), 100 mm long, anchored by two verbal descriptors (0 mm being the total absence of pain and 100 mm being the worst imaginable pain). The measurement of the average change in the intensity of NP (baseline) will be performed by comparing the value on the first visit (day 0) with the value on the final visit (day 56).
Incidence of Serious Treatment-Emergent Adverse Events assessed by a questionnaire | 56 days
  The Incidence of Serious Treatment-Emergent Adverse Events will be assessed by measuring the number of participants who experience Serious Adverse Events with the use of methadone or placebo. The search for the adverse events will be done with a questionnaire containing the main adverse events previously described in the medical literature and in the manufacturer's label (methadone). In addition, unexpected adverse events will also be described in detail and reported to the responsible institution. The definition of a serious treatment adverse event will be made in accordance with the rules of the National System of Notifications for Health Surveillance-NOTIVISA. Each serious adverse event will be described in detail and notified to the responsible institution.The comparison between the incidence of Serious Treatment-Emergent Adverse Events will be made between the groups (methadone and placebo) at the end of the study.
Incidence of methadone addiction/misuse or withdrawal syndrome assessed by a prespecified questionnaire | 56 days
  The incidence of methadone addiction/misuse or withdrawal syndrome will be assessed by a prespecified questionnaire, containing eight clinical characteristics that may be related to the methadone addition/misuse or withdrawal syndromes. If one or more of those 8 characteristics listed in the questionnaire are present, an immediate communication will be made to the assistant physician (for diagnostic confirmation and referral to multidisciplinary treatment), as well as the exclusion of the individual from the study (after discussion with the research coordinators).

SECONDARY OUTCOMES:
Incidence of drop-outs due to Non-Serious Treatment-Emergent Adverse Events assessed by a questionnaire | 56 days
  The incidence of Non-Serious Treatment-Emergent Adverse Events will be assessed (at the end of the study) measuring the proportion of participants who experienced non-serious adverse events in each study group and the proportion of drop-out losses caused by such effects.The search for the adverse events will be done with a questionnaire containing the main adverse events previously described in the medical literature and in the manufacturer's label (methadone). In addition, unexpected adverse events will also be described in detail and reported to the responsible institution.

OTHER OUTCOMES:
Improvement in sleep quality, assessed by The Medical Outcomes Study Sleep Problem Index II (SPI II) | 56 days
  It will be investigated whether there is a correlation between the use of Methadone and the improvement of sleep quality in relation to placebo. The MOS questionnaire, frequently used in chronic pain syndromes, is composed of 12 questions about the main aspects of sleep, evaluated through a categorical scale (from 1: permanent, to 6: never). The nine items of the Medical Outcomes Study Sleep Problem Index II (SPI II) are part of the 12-item Medical Outcomes Study Sleep Scale, with a final score ranging from 0 to 100, with higher scores indicating more sleep problems. The main target would be to reduce the SPI II score by at least 10 points with the use of methadone.
Improvement in mood and anxiety symptoms, assessed by The Hospital Anxiety and Depression Scale (HADS) | 56 days
  It will be evaluated whether there is a correlation between the use of Methadone and the improvement of symptoms of Depression and/or Anxiety (in those patients who may have these symptoms prior to the beginning of the study) in relation to placebo. The HADS questionnaire allows assessing, over a week, on a scale from 0 to 3, the intensity of symptoms of anxiety or depression. It consists of 7 questions to assess anxiety and 7 questions to assess depression, each one (depression or anxiety) being evaluated on a maximum scale of 21 points. A score equal to or greater than 8 on the HADS for either anxiety or depression suggests a significant impact.
Improvement in quality of life, assessed by The Short-Form 6 dimensions Questionnaire (SF-6D) | 56 days
  It will be researched if there is a correlation between the use of Methadone and the improvement in the quality of life of patients in relation to placebo. The SF-6D is a quality of life self-assessment questionnaire that allows for obtaining measures of preference for health states. It has 6 health dimensions (functional capacity, physical and emotional aspects, social aspects, pain, mental health and vitality) with 4-6 levels each. The SF-6D score, which ranges from 0 to 1, represents the strength of an individual's preference for a particular health state, on a scale where 0 is equal to the worst health state and 1 means the best health state. The total SF-6D value is the summation of 6 dimensions scoring.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C. de Andrade, PhD, Study Chair — University of Sao Paulo
Locations (1):
- University of São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The complete IPD will be shared with other authors who wish to use it in individual patient data (IPD) meta-analysis. Other specific situations will be discussed on a case-by-case basis.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD will be available after the estimated study completion time (August/2021) and for five years.
Access Criteria: The complete IPD will be sent by e-mail after other researchers request it for use in individual patient data (IPD) meta-analysis. Other specific situations will be discussed on a case-by-case basis.

REFERENCES:
- [Derived] Pentiado Junior JAM, Barbosa MM, Kubota GT, Martins PN, Moreira LI, Fernandes AM, da Silva VA, Junior JR, Yeng LT, Teixeira MJ, Ciampi de Andrade D. METHA-NeP: effectiveness and safety of methadone for neuropathic pain: a controlled randomized trial. Pain. 2025 Mar 1;166(3):557-570. doi: 10.1097/j.pain.0000000000003413. Epub 2024 Oct 22. PMID 39432734